CLINICAL TRIAL: NCT00017706
Title: Treatment of Obesity in the Primary Care Setting
Brief Title: Effectiveness of Primary Care Physicians in Delivering Weight Control Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: Simkin-Silverman (completed); DK52050
Record Dates: First submitted 2001-06-07; First posted 2001-06-07 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: physician education; behavioral weight control; physician intervention; obesity counseling
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: physician-delivered weight control

SUMMARY:
This randomized clinical trial will determine the efficacy of physicians providing weight control advice to their overweight and obese patients in primary care practice.

DETAILED DESCRIPTION:
Enrolled physicians are randomly assigned to receive brief training in either: 1) behavioral weight control intervention or 2) obesity education. Enrolled patients are asked to see their physician for 2 weight control consultations during the year to discuss their weight and physical activity. Regardless of the training the physician receives, the weight control advice is tailored to the individual patient. Patients include men and women between the ages of 21 - 70 years, with a Body-Mass Index of 27 or greater, and they have met medical and other study eligibility criteria in order to safely participate. As a participant in the trial, all patients are asked to attend an initial baseline assessment, and two follow-up assessments; 3 and 12 months after their first weight control consultation visit with their physician in order to evaluate any changes in their weight, waist circumference, physical activity, eating patterns, and mood. The findings of this important study will shed light upon the role physician advice may have in helping overweight and obese patients lose weight and become more physically active.

ELIGIBILITY:
Inclusion Criteria:

* Body-Mass Index greater than or equal to 27
* Able to walk without assistance
* No untreated hypothyroidism or Cushing Disease
* No unstable medical or psychiatric condition
* No signs or symptoms of cardiovascular disease
* No history of gallstones
* No terminal illness
* No other acute or chronic medical condition in which weight loss is contraindicated
* Medically cleared for physical activity

Exclusion Criteria:

* Pregnant, nursing or planning to become pregnant in the next year
* Had an in-patient hospital stay in the last 3 months
* Lost more than 10 lbs in the last 4 months
* Taking an OTC or prescribed medication for weight loss
* In treatment for an eating disorder
* In treatment for depression (if patient is on an anti-depressant and has not had a recent episode of depression in the past 3 months then he/she is eligible)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2001-05

CONTACTS AND LOCATIONS:
Overall Officials: Laurey Simkin-Silverman, Ph.D., Principal Investigator — University of Pittsburgh, GSPH, Department of Epidemiology
Locations (1):
- University of Pittsburgh, GSPH, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Simkin-Silverman LR, Wing RR. Management of obesity in primary care. Obes Res. 1997 Nov;5(6):603-12. doi: 10.1002/j.1550-8528.1997.tb00582.x. PMID 9449146